CLINICAL TRIAL: NCT03127930
Title: Improving Caregiver Mediated Medication Management
Brief Title: Improving Caregiver Mediated Medication Management- The 3M Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Judith Erlen, Professor of Nursing, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO08050015
Record Dates: First submitted 2017-04-18; First posted 2017-04-25 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Medication Management
Keywords: Cognitive Impairment; Memory loss; Caregivers; Medication adherence; Medication compliance; Medication management; Problem solving; Quality of Life; Health resource utilization; Community dwelling
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders; Medication Adherence | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Social Cognitive and Self Efficacy Theory drove the problem-solving tailored intervention delivered via face to face and telephone by either a master's prepared social worker or nurse.
Who Masked: Investigator
Masking Description: Participants and outcomes assessors were not blind to the intervention by nature o the protocol. Investigators and analysts were blinded to study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention: Participants receive both usual care including a standard brochure on patient management provided by the Alzheimer's Association plus a tailored problem-solving intervention to improve caregiver's management of medications for their family or friend care recipient who has memory deficit.
  Interventions: Behavioral: Intervention
- Usual Care (No Intervention): No Intervention: Participants do not receive the problem solving intervention and are followed as a Usual Care condition including receiving a standard brochure on patient management provided by the Alzheimer's Association. .

INTERVENTIONS:
Behavioral: Intervention — Participants receive 5 individualized contacts (home visits and phone calls) with either a social worker or a nurse to develop problem solving skills as applied to medication management.
  Other Names: Problem Solving training to improve medication management
  Arms: Intervention

SUMMARY:
This study sought to improve medication management by caregivers of community dwelling patients with dementia or simple memory loss. This was done by testing a tailored intervention delivered both in-home and by telephone by either a social worker or nurse. The intervention was designed to decrease medication deficiencies and improve medication adherence by developing problem solving skills.

DETAILED DESCRIPTION:
Objective: The overall purpose of this investigation is to test the efficacy of a tailored caregiver mediated medication management intervention designed for caregivers of community dwelling patients with dementia.

Specific Aims:

Primary Aim:

Examine the efficacy of a tailored caregiver mediated medication management in-home and telephone delivered intervention designed to decrease medication taking deficiencies and daily hassles and improve medication adherence of caregivers of community dwelling patients with dementia vs. standard education/usual care group of caregivers over time.

Hypothesis 1 Immediately post-treatment (8 weeks), there will be a decrease in medication taking deficiencies and daily hassles and an improvement in caregiver medication adherence in the treatment compared to the usual care group.

Hypothesis 2 Immediately post-maintenance (16 weeks), there will be a sustained decrease in medication taking deficiencies and daily hassles and an improvement in caregiver medication adherence in the treatment group compared to the usual care group.

Hypothesis 3 At 8 weeks post-maintenance (24 weeks), there will continue to be a sustained decrease in medication taking deficiencies and daily hassles and an improvement in caregiver medication adherence in the treatment group compared to the usual care group.

Secondary Aims:

1. Examine the efficacy of a tailored caregiver mediated medication management in-home and telephone delivered intervention designed to decrease medication taking deficiencies and daily hassles and increase medication adherence of caregivers of community dwelling patients with dementia vs. standard education/usual care group of caregivers on the distal outcome of adverse patient outcomes including unplanned doctor's visits, emergency room visits, and hospitalizations over time.
2. Examine the efficacy of a tailored caregiver mediated medication management in-home and telephone delivered intervention designed to decrease medication taking and daily hassles and increase medication adherence of caregivers of community dwelling patients with dementia vs. standard education/usual care group of caregivers on the distal outcome of health related quality of life in both caregivers and community dwelling patients over time.

Significance: This study is both timely and significant because of the growing number of patients with dementia who need supportive services of family members, as well as from the health care system. This study is addressing a very timely issue, the reduction of medication deficiencies that can lead to errors. This is a priority patient safety issue regardless of whether the medications are given by a professional healthcare provider or an informal family caregiver. Additionally, this intervention has the potential for translation into geriatric practices and lay community or support groups.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS 18 years of age or older; Patient having memory deficit reported by either member of dyad. Be unable to manage their own medications Have a minimum of two co-morbid conditions (one additional condition besides dementia) Have more than one medication prescribed or recommended by an MD. This could include MD recommended supplements and over the counter medications.

Have an informal caregiver/not a paid caregiver; Live within approximately a 75 mile radius of the University of Pittsburgh.

INFORMAL/FAMILY CAREGIVERS 18 years of age or older; have access to a telephone for the telephone-delivered intervention and maintenance sessions; have medication management deficiencies as identified by the Medication Management Instrument for Deficiencies on the Elderly (MedMaIDE) at screening; live within a 75 mile radius of the University of Pittsburgh.

-

Exclusion Criteria:

PATIENTS:

major physical/aggressive behavior problems identified at screening using the Revised Memory Behavior Problem Checklist.

INFORMAL/FAMILY CAREGIVERS:

hearing impairment without a modified telephone to enhance their ability to hear.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2013-07-30 (Actual); Study Completion 2013-07-30 (Actual)

PRIMARY OUTCOMES:
Medication management assessed by investigator developed Medication Deficiency Checklist- post-treatment | 8 weeks
  Improved medication management of patient's medications by caregiver at post-intervention.
Medication management-assessed by investigator developed Medication Deficiency Checklist- post maintenance | 16 weeks
  Maintenance of improved medication management of patient's medications by caregiver following a booster/maintenance period
Medication management-assessed by investigator developed Medication Deficiency Checklist- post followup | 24 weeks
  Maintenance of improved medication management of patient's medications by caregiver after a no treatment followup period.

SECONDARY OUTCOMES:
Patient outcomes- medical utilization-Investigator developed Unscheduled Event Checklist | 24 weeks
  decrease medical utilization such as md visits, emergency visits, and hospitalizations
Caregiver outcome- Improved quality of life via Medical Outcome Short Form (SF-36) | 24 weeks
  Improvement of caregiver's quality of life over time

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Erlen, RN, PhD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erlen JA, Lingler J, Sereika SM, Tamres LK, Happ MB, Tang F. Characterizing caregiver-mediated medication management in patients with memory loss. J Gerontol Nurs. 2013 Apr;39(4):30-9. doi: 10.3928/00989134-20130220-91. Epub 2013 Feb 28. PMID 23445184
- [Result] Lingler JH, Sereika SM, Amspaugh CM, Arida JA, Happ ME, Houze MP, Kaufman RR, Knox ML, Tamres LK, Tang F, Erlen JA. An intervention to maximize medication management by caregivers of persons with memory loss: Intervention overview and two-month outcomes. Geriatr Nurs. 2016 May-Jun;37(3):186-91. doi: 10.1016/j.gerinurse.2015.12.002. Epub 2016 Jan 21. PMID 26804450
- [Result] Tang F, Jang H, Lingler J, Tamres LK, Erlen JA. Stressors and Caregivers' Depression: Multiple Mediators of Self-Efficacy, Social Support, and Problem-Solving Skill. Soc Work Health Care. 2015;54(7):651-68. doi: 10.1080/00981389.2015.1054058. PMID 26317766